CLINICAL TRIAL: NCT02036840
Title: Perioperative Antibiotic Choices for Surgical Prophylaxis in Penicillin-allergic Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chairman - Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB11-00822
Record Dates: First submitted 2014-01-13; First posted 2014-01-15 (Estimated); Results first posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Penicillin Allergy
MeSH Terms: interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Penicillin allergy
  Interventions: Drug: Antibiotic

INTERVENTIONS:
Drug: Antibiotic

SUMMARY:
The proposed research project will retrospectively review the anesthetic records over the past 5 years and identify patients who present with a history of penicillin allergy or allergy to an antibiotic in the penicillin family. The reason for that history and the facts on which that allergy are noted will be determined. Additionally, the choice of antibiotic prophylaxis will be recorded and any adverse effect to that antibiotic noted. We will also note whether appropriate timing of the antibiotic is achieved.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are labeled as penicillin or penicillin family allergic.

Exclusion Criteria:

* As neurosurgical patients routinely receive vancomycin at NCH for surgical prophylaxis, they will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a history of allergy to penicillin who required antibiotic prophylaxis prior to/during surgery.
Sampling Method: Non-Probability Sample
Enrollment: 513 (Actual)
Dates: Start 2013-01; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Penicillin Allergy: Antibiotic
Period: Overall Study
Arm/Group | Penicillin Allergy
Started | 513
Completed | 513
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Penicillin Allergy
Number analyzed (Participants) | 513
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 513
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250
  Male | 263
Region of Enrollment [Number; unit: participants]
  United States | 513

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Antibiotic Related Adverse Event
Time Frame: 24 hours
Measure: Number; unit: participants
Arm/Group | Penicillin Allergy
Number analyzed (Participants) | 513
participants | 12

ADVERSE EVENTS:
Description: Please note: This is a retrospective chart review so the antibiotic related adverse events listed below occurred before the study even started.
Arm/Group | Penicillin Allergy
Serious Adverse Events (participants affected / at risk) | 0/513
Other Adverse Events (participants affected / at risk) | 12/513
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Penicillin Allergy (N=513)
Hives (Immune system disorders) | 4
Erythema (Immune system disorders) | 1
Rash (Immune system disorders) | 6
Hypotension (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes